CLINICAL TRIAL: NCT01438775
Title: Phase 3 Multicenter Prospective Open Label Clinical Safety Evaluation of Re-Injection of NX-1207 for the Treatment of BPH: Two Doses 1-7 Years Apart
Brief Title: Phase 3 Evaluation of Re-Injection of NX-1207 for the Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX02-0020
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH; Enlarged prostate; Lower urinary tract symptoms; LUTS; LUTS secondary to BPH; LUTS/BPH; Benign prostatic obstruction; BPO; Bladder outlet obstruction; BOO
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction | interventions — fexapotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Injection of NX-1207 (Experimental): Intraprostatic injection of 2.5 mg NX-1207
  Interventions: Drug: NX-1207

INTERVENTIONS:
Drug: NX-1207 — 2.5 mg NX-1207 in 10 mL saline vehicle

SUMMARY:
This study is designed to demonstrate the safety and efficacy of a second transrectal intraprostatic injection of NX-1207 given to subjects with Benign Prostatic Hyperplasia (BPH) who previously received an injection of NX-1207 in an earlier U.S. clinical trial of NX-1207.

ELIGIBILITY:
Inclusion Criteria:

* Be male aged 45 or older.
* Sign an informed consent form.
* Be in good health.
* Received NX-1207 in a previous completed study or received NX-1207 or placebo in a concurrent U.S. study (NX02-0017 and NX02-0018) and completed their V10 (365 day) visit.
* Have Prostate Gland Volume ≥ 25 mL (25 g).

Exclusion Criteria:

* Surgery or minimally invasive surgical therapy (MIST) for treatment of BPH after first NX-1207 injection
* Post-void residual urine volume > 200 mL
* Presence of a symptomatic median lobe of the prostate
* History of use of self-catheterization for urinary retention.
* Urinary retention in the previous 12 months.
* Prostatitis
* Urinary tract infection more than once in the past 12 months
* Prostate or bladder cancer.
* PSA ≥10 ng/mL
* Poorly controlled diabetes
* History or evidence of illness or condition that may interfere with study or endanger subject
* Participation in a study of any investigational drug (other than NX-1207) or investigational device within the previous 90 days
* Use of specific prescribed medications that may interfere with study or endanger subject

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety | 180 days
  Safety parameters as determined by Adverse Events, clinical laboratory test results, vital signs, physical exam and electrocardiogram (ECG).

SECONDARY OUTCOMES:
Symptomatic Improvement | 90 days
  Symptomatic improvement as measured by the change in American Urological Association (AUA) Symptom Index from baseline at 90 days. The AUA Symptom Index is a standardized questionnaire that uses seven questions relating to associated BPH symptoms to provide an assessment of symptom severity on a scale from 0 (no symptoms) to 35 (most severe).
Prostate Volume Change | 90 days
  Change in prostate volume from baseline to 90 days as measured by transrectal ultrasonography
Change in Urinary Peak Flow | 90 days
  Change in Urinary Peak Flow (Qmax) from baseline to 90 days as determined by urinary flow-rate recording (uroflowmetry).
Symptomatic Improvement | 180 days
  Symptomatic improvement as measured by the change in AUA Symptom Index from baseline at 180 days.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Huntsville, Alabama
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Atherton, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., San Diego, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Tarzana, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Denver, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Englewood, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New Britain, Connecticut
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Sarasota, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Meridian, Idaho
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Forest Hill, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Jeffersonville, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Shreveport, Louisiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Annapolis, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Southaven, Mississippi
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Missoula, Montana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Lawrenceville, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Albuquerque, New Mexico
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Brooklyn, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Garden City, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New York, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Poughkeepsie, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Concord, North Carolina
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Bismarck, North Dakota
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Lancaster, Pennsylvania
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Memphis, Tennessee
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Arlington, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Houston, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, San Antonio, Texas